CLINICAL TRIAL: NCT03448796
Title: High Tibial Opening Wedge Osteotomy and Conservative Treatment in Medial Knee Osteoarthritis - A Randomised Controlled Trial
Brief Title: Opening Wedge High Tibial Osteotomy
Acronym: OHTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with recruiting patients.
Sponsor: Kuopio University Hospital (Other)
Collaborators: Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5203099
Record Dates: First submitted 2017-03-02; First posted 2018-02-28 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthrosis of Knee; Osteoarthritis, Knee
Keywords: High tibial osteotomy; Osteoarthrosis; Tomofix; Randomized controlled trial
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The clinical assessors are blinded when applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HTO-group (Active Comparator): Group receives opening wedge high tibial osteotomy with Tomofix -plate. Operative intervention is followed by supervised physiotherapeutic rehabilitation.
  Interventions: Procedure: HTO; Other: Supervised physiotherapeutic program
- FT -group (Active Comparator): Group receives only supervised physiotherapeutic rehabilitation.
  Interventions: Other: Supervised physiotherapeutic program

INTERVENTIONS:
Procedure: HTO — Group that receives high tibial osteotomy combined with supervised physiotherapy as treatment.
  Arms: HTO-group
Other: Supervised physiotherapeutic program — Group that receives only supervised physiotherapy as treatment.

SUMMARY:
A prospective, randomised controlled trial where clinical and radiological outcome of high tibial opening wedge osteotomy with physiotherapy is compared to physiotherapy alone while treating symptomatic medial knee osteoarthrosis.

DETAILED DESCRIPTION:
90 Symptomatic patients with mild to moderate medial knee osteoarthrosis are randomized to two groups:

Group 1 (HTO-group) receive an diagnostic arthroscopy with high tibial opening wedge osteotomy (Tomofix-plate). Postoperatively a supervised physiotherapeutic rehabilitation program is started.

Group 2 (FT-group) receive the same supervised physiotherapeutic rehabilitation program without the HTO or arthroscopy.

Primary outcome measure is composite score of Knee injury and Osteoarthritis Outcome Score (KOOS5).

Secondary outcome measures are pain (VAS), KOOS subscales, objective physical performance measurements, progression of osteoarthrosis (X-ray, MRI), change of mechanical axis, complications, treatment costs, rate of reoperation, revision to total knee arthroplasty (TKA), biological markers of arthrosis progression, 15D (quality of life assessment), QALY (Quality-Adjusted Life-Year), Work Productivity and Activity Impairment Questionnaire, Work Productivity and Activity Impairment Questionnaire, sum of governmental benefits received.

Outcomes will be measured at 24, 60 and 120 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pain: Subjective pain in the knee most of the month for at least one month during past 12 months.
* Knee range of motion (ROM) at least 5-120 degrees
* X-ray: medial joint space Altman > 1. Lateral joint space Altman < 2.
* Mechanical axis > 3 degrees varus alignment.
* Medial proximal tibial angle (MPTA) < 90 degrees
* age 25-55.
* Written consent, accepts both treatment arms.

Exclusion Criteria:

* Pain is caused by something else than medial knee osteoarthrosis
* deficient ROM (flexion contracture > 10 degrees, flexion < 110 degrees)
* significant ligament instability
* post traumatic OA
* clinically relevant neurological disease (e.g. Alzheimer´s disease)
* clinically relevant metabolical disease (e.g. Diabetes)
* alcohol/drug abuse
* infectious/inflammatory joint disease
* previous knee area osteotomy or lower limb arthroplasty
* smoking (> 0 cigarette per day)
* obesity (BMI > 33)
* pregnancy or hope of pregnancy in the following two years

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Change of KOOS5 | 24, 60, 120 months
  The change of Composite score of Knee injury and Osteoarthritis Outcome Score (KOOS) subscales

SECONDARY OUTCOMES:
Change of pain measured in numeric rated scale (NRS) | 24, 60, 120 months
  Amount of subjective (knee) pain
Change of KOOS subscales | 24, 60, 120 months
  Individual subscales of Knee injury and Osteoarthritis Outcome Scores
Change in results of 40 meter fast paced walk test | 24, 60, 120 months
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft)
Change in results of stair climb test | 24, 60, 120 months
  The time (in seconds) it takes to ascend and descend a flight of stairs
Change in results of timed up and go test | 24, 60, 120 months
  Time (seconds) taken to rise from a chair, walk 3 m, turn, walk back to the chair, then sit down wearing regular footwear and using a walking aid if required.
Radiological progression of arthrosis | 24, 60, 120 months
  x-ray, MRI
Change in mechanical axis of lower limb | 12, 24, 60, 120 months
  As measured from whole leg standing radiograph
Incidence of complications | Up to 120 months
  eg infection, non-union, thromboembolic complications etc.
Total costs of treatment | Up to 120 months
  Including the cost of hospital treatment, physiotherapy, cost of medication, cost of sick leave
Incidence of reoperation | Up to 120 months
  Amount of reoperations needed
Hyaluronic acid (HA) concentration | 24, 60, 120 months
  At 24, 60 and 120 month follow-up blood and synovial fluid samples are analyzed for HA concentration.
  This will be measured with antibody-ELISA at mg/g from 10µl of fluid. The same measurement will be conducted on blood serum.
Fatty acid (FA) profiling | 24, 60, 120 months
  At 24, 60 and 120 month follow-up blood and synovial fluid samples are analyzed for fatty acid (FA) profiling. FA will be analyzed from 75 µl of synovial fluid and 200 µl of blood serum with gas chromatography as mol-%.
Synovial fluid composition | 24, 60, 120 months
  At 24, 60 and 120 month follow-up synovial fluid samples are analyzed for composition.
  Synovial fluid composition will be assessed visually with confocal microscopy with a HA-biding fluorescent probe and Nile red probe that show both HA particles and the association of these particles on extracellular vesicles to assess the significance of vesicle-mediated HA secretion into synovial fluid.
General variables reflecting inflammatory status | 24, 60, 120 months
  At 24, 60 and 120 month follow-up blood and blood serum samples are analyzed for general variables reflecting inflammatory status (leucocytes, C-reactive protein, IL-6).
15D -quality of life assessement | 24, 60, 120 months
  The change of health-related quality of life (HRQoL) instrument
Work Productivity and Activity Impairment Questionnaire (WPAI) | 24, 60, 120 months
  The change of WPAI
Amount of national benefits received | Up to 120 months
  The amount of benefits are gathered from:
  1. The hospital discharge register (maintained by National Institute for Health and Welfare)
  2. National benefits paid by The Social Insurance Institution of Finland
  3. Pension decision made by Finnish Centre for Pensions

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Jalkanen, M.D., Principal Investigator — Kuopio University Hospital
Locations (1):
- University Hospital of Kuopio, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Undecided